CLINICAL TRIAL: NCT05819814
Title: Polygenic Risk-based Detection of Subclinical Coronary Atherosclerosis and Change in Cardiovascular Health
Acronym: PROACT 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Akl C. Fahed, MD, MPH, Interventional Cardiologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023P000935
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Polygenic risk score; Genetics; Genomic medicine; Precision medicine; Preventive cardiology; Risk prediction; Cardiovascular health; Coronary CT angiogram; Coronary plaque; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Genetic Risk Score; Atherosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants will receive their high polygenic risk result for coronary artery disease.
  Interventions: Genetic: Disclosure of high polygenic risk result for coronary artery disease
- Control (No Intervention): Participants will receive standard of care, and disclosure of high polygenic risk result will be deferred until study completion.

INTERVENTIONS:
Genetic: Disclosure of high polygenic risk result for coronary artery disease — The disclosure of a high polygenic risk result for coronary artery disease involves a clinical report coupled with a virtual meeting with a genetic counselor.
  Arms: Intervention

SUMMARY:
The goal of this randomized controlled trial is to assess the impact of disclosing a high polygenic risk result for coronary artery disease on change in cardiovascular health over one year.

DETAILED DESCRIPTION:
The main question PROACT 1 aims to answer is whether cardiovascular health improves following disclosure of high polygenic risk result for coronary artery disease compared to standard of care.

This is a 1:1 randomized controlled trial of middle-aged participants with no known cardiovascular disease, are not on lipid-lowering therapy, who have high polygenic risk score for coronary artery disease, and do not have quantifiable plaque on coronary computed tomography angiography. Participants will be randomized into two equal groups: one group will receive their high polygenic risk result for coronary artery disease at baseline, and the other group will receive their result after study completion at 1 year. Change in cardiovascular health as measured by the American Heart Association Life's Essential 8 score from baseline to one-year will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 40 and 75 years of age capable and willing to provide informed consent
* Participant has high CAD PRS as defined on a clinical test

Exclusion Criteria:

* Participant with a history of cardiovascular disease, defined by a diagnosis of coronary artery disease, peripheral artery disease, or cerebrovascular disease
* Participant with quantifiable plaque on a coronary computed tomography angiography
* Participant with a history of Liver disease (cirrhosis, active hepatitis, or severe hepatic disease) or any of the following recent lab results and determined to be non-transient: alanine aminotransferase greater than 3 times the upper limit of normal or total bilirubin greater than 2 times the upper limit of normal (unless due to Gilbert syndrome)
* Participant with estimated glomerular filtration rate <60 mL/min/1.73 m2 or creatinine greater than 2 times the upper limit of normal
* Patient with history of an allergic reaction or significant sensitivity to iodinated contrast, colchicine, or statins
* Patient currently taking LDL cholesterol lowering or anti- inflammatory medications including colchicine
* Participants requiring regular drugs known to be potent CY2P inhibitors (eg. ketoconazole, clarithromycin)
* Female patient who is pregnant, or breast-feeding or is considering becoming pregnant during the study
* Participant with BMI ≥ 40 kg/m2
* Participant unable to provide informed consent
* Participant unable to hold breath for 10 seconds

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Assess the impact of disclosing a high polygenic risk result for coronary artery disease on change in cardiovascular health | 1 year
  Change in cardiovascular health from baseline to one year as measured by the American Heart Association's Life's Essential 8 (LE8) Score will be compared between an intervention arm that receives a high polygenic risk result for coronary artery disease and a control group that receives standard of care. The LE8 score ranges between 0 and 100 with higher numbers indicating better cardiovascular health.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No